CLINICAL TRIAL: NCT04068506
Title: Comparison of Analgesic Effects of Gabapentin and Paracetamol in Patients With Hand Injury
Brief Title: Analgesic Effects of Gabapentin and Paracetamol
Acronym: GABA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hyder Ali, assistant professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 123
Record Dates: First submitted 2018-11-11; First posted 2019-08-28 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Hand Injuries
MeSH Terms: conditions — Hand Injuries | interventions — Gabapentin

STUDY DESIGN:
Intervention Model Description: A total of 50 patients who fulfill the inclusion criteria will be approached and written consent will be signed by the participants prior to the interview. Participants will be divided into two groups divided equally i.e. gabapentin group and paracetamol group. Gabapentin group received 600 mg dose while the control/other group received 1 gram (1000 mg) of paracetamol as a postoperative analgesic agent.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators will divide the calculated sample size into two groups A and B in which all the participants have the same probability of being included in the study. Two unrecognizable envelopes separating both drugs gabapentin and paracetamol with equivalent dose will be administered with the specific code number labeled by the principal investigator and will be prescribed by the on-duty doctor to the patients in tablet form once orally allowed after surgery. Analgesic effects will be inquired after 6 hours of drug administration. Further questions will be asked according to the questionnaire by the co-investigators having no knowledge of the given drug to participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Gabapentin 600 mg Tab
  Interventions: Drug: Gabapentin 600 mg Tab
- Group B (Active Comparator): Paracetamol 1000 mg Tab
  Interventions: Drug: Gabapentin 600 mg Tab

INTERVENTIONS:
Drug: Gabapentin 600 mg Tab — Gabapentin 600 mg Tab is a drug of choice for treating postoperative pain.
  Other Names: Neurontin

SUMMARY:
This research is about the effects of drug gabapentin; which is an amino acid that is structurally similar to neurotransmitter GABA. It is a novel drug used for the treatment of postoperative pain with analgesic properties having unique mechanism of action. This study reviews clinical effects of this agent in hand injury patients managed at the Department of Plastics & Reconstructive Surgery, Dow University of Health Sciences & Dr. Ruth KM Pfau Civil Hospital Karachi.

This study aims to inquire the analgesic properties of gabapentin in the patients and to further investigate its comparison with the equivalent dose of paracetamol given 6 hours after undergoing operative procedure. Acetaminophen is well tolerated when administered in therapeutic dose for pain management. It is a principal drug used as pain reliever and as an antipyretic regimen.

This is an experimental study in which a pre-coded questionnaire would be approved in the research for appraising the intensity of pain after intervening operative procedure using visual analogue scale, measuring the pain intensity from 0-10. The questions regarding pain intensity will be inquired after administrating the drug six hours postoperatively. The drug will be prescribed by the doctor on duty having no knowledge regarding the given drug or the group in which he/she is administrating the drug; further questionnaire will be filled by the two co-investigators who will be trained by principal investigator, how to take correct information.

Sample size was calculated using www.openepi.com using the previous literature searches of similar research and 50 patients (25 in each group) will be randomly selected from the ward of a known case of hand injury. Group A patients will receive 600 mg of gabapentin post operatively while group B will receive 1 g of paracetamol for management of pain postoperatively orally.

DETAILED DESCRIPTION:
Gabapentin is an anti-convulsion medication and has a high affinity for voltage-gated calcium channel throughout the brain, acts by inhibition of release of excitatory neurotransmitters. As a lipophilic substance, it shows linear pharmacokinetics and has oral bioavailability greater than 90%. Gabapentin is used in a variety of condition as a therapeutic measure involving diabetic neuropathy, post-herpetic neuralgia, in partial seizures, restless leg syndrome, post-menopausal hot flashes, anxiety, resistant mood disorders, essential tremors, and numerous other modalities. Gabapentin is a muscle relaxant and anti-spasmodic, its analgesic effect has also be identified for moderate to severe pain.

ELIGIBILITY:
1. Inclusion Criteria:

   1. Patients between 18-60 years of age
   2. Patients Undergoing hand surgery in the Department of Plastics and Reconstructive Surgery, Dr. Ruth KM Pfau Civil Hospital Karachi, Dow University of Health Sciences
2. Exclusion criteria:

   1. Pregnant women
   2. Any patient presenting with the signs of:

      * Arrhythmia
      * Myocardial ischemia
      * Cognitive impairment
      * Psychiatric disorders
      * Drug abuse
   3. Patients sensitive to any epileptic drug or taking any anti-epileptic drug
   4. Having severe and multiple injuries.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Comparison of analgesic effects of Gabapentin and paracetamol in patients with hand injury | 6 months
  The outcome of this study will be finding that how much gabapentin is effective in improving pain over paracetamol by simply inquiring about the analgesic effect of both drugs with the help of Visual analogue scale measuring pain intensity from 1 - 10 and how much each drug adversely effects individual's health by assessment of any unwanted symptoms like: nausea, vomiting, headache, dizziness, etc. So, that certainty about its effect and efficacy over paracetamol in relieving pain can be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Hyder Ali, MBBS,FCPS, Principal Investigator — Assistant professor at Dr.Ruth K.M pfau Civil Hospital Karachi,DUHS
Locations (1):
- Dr. Ruth K.M. Pfau Civil Hospital Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ali H; Naveed; Perveen B. Comparison of analgesic effects of Gabapentin and Paracetamol post-operatively in patients with hand injury. J Pak Med Assoc. 2021 Nov;71(11):2501-2505. doi: 10.47391/JPMA.359. PMID 34783725
- See also: Improving the Quality of Care Through Pain Assessment and Management. — https://www.ncbi.nlm.nih.gov/books/NBK2658/
- See also: A descriptive study of hand injuries presenting to the adult emergency department of a tertiary care center in urban India. — http://www.onlinejets.org/article.asp?issn=0974-2700;year=2017;volume=10;issue=1;spage=19;epage=25;aulast=Ghiya
- See also: Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. — https://www.ncbi.nlm.nih.gov/pubmed/12873949
- See also: Gabapentin in Acute Postoperative Pain Management — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4009126/
- See also: Pain as a factor complicating recovery and discharge after ambulatory surgery. — https://www.ncbi.nlm.nih.gov/pubmed/12198050
- See also: Prescribing gabapentin off label: Perspectives from psychiatry, pain and neurology specialists — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3567599/
- See also: Randomized, controlled, multicentre clinical trial of the antipyretic effect of intravenous paracetamol in patients admitted to hospital with infection — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5346867/